CLINICAL TRIAL: NCT00202189
Title: Acute Effects of Inhaled Corticosteroids on Dynamic Airway Function During Rest and Exercise in Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Effects of Inhaled Corticosteroids in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Dr. Denis O'Donnell, Queen's University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: DMED-892-05
Record Dates: First submitted 2005-09-09; First posted 2005-09-20 (Estimated); Last update posted 2008-08-13 (Estimated); Status verified 2008-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Pulmicort; Budesonide; Chronic; Obstructive; Pulmonary; Disease; Exercise; Emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchiolitis Obliterans Syndrome; Disease; Motor Activity; Emphysema | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Budesonide
  Interventions: Drug: Budesonide
- 2 (Placebo Comparator): Saline Solution (0.9% NaCl)
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: Budesonide — Nebulized Budesonide (4 mL) or saline solution (0.9% NaCl) (4 mL) will be administered to subjects once only.
  Other Names: Pulmicort

SUMMARY:
Human and animal studies have shown that inhaled corticosteroids (ICS) decrease airway blood flow . This effect is immediate (within 30 minutes), transient (lasting 90 minutes), and in animal studies independent of gene expression. In COPD patients, decrease in bronchial blood flow may also decrease mucosal edema, airway resistance and improve small airway function. If such an effect exists, then we should be able to measure improvements in airway conductance and reduce lung hyperinflation, which would have salutary effects on dyspnea and exercise endurance.

To our knowledge, no study has examined the immediate effect of ICS on small airway function in COPD. The purpose of this study is to examine the effects of nebulized Pulmicort on small airway function (spirometry, plethysmographic lung volumes, airways resistance, closing volume, partial flow-volume loop analysis) and exercise endurance in patients with moderate to severe COPD.

HYPOTHESIS

1. Nebulized ICS will immediately improve airway function compared with placebo (nebulized saline).
2. Enhanced lung emptying and reduced operating lung volumes during rest and exercise following ICS therapy will translate acutely into clinically important reductions in exertional dyspnea and improvements in exercise endurance.

DETAILED DESCRIPTION:
This will be a single site, pilot, randomized, double-blinded, placebo-controlled, cross-over study that will be conducted at this centre. Subjects will be required to complete four (4) visits to the laboratory over a one-month period.

At Visit 1, subjects who meet all study inclusion and exclusion criteria, will have a full set of pulmonary function tests (PFT) done and complete a symptom-limited incremental cycle exercise test. At Visit 2, subjects will have a partial set of pulmonary function tests (PFT) done and complete a symptom-limited constant load cycle exercise test. On the third and fourth visit subjects will be randomized to treatment with either nebulized saline or nebulized Pulmicort® in a double blinded, cross-over design, subsequent to which they will have their PFT's and symptom limited constant load exercise testing done.

ELIGIBILITY:
Inclusion Criteria:

* FEV1 less than/equal to 70 % predicted, FEV1/FVC ratio less than/equal to 70%, and FRC greater than/equal to 120 % predicted
* Moderate to severe chronic activity-related dyspnea (modified Baseline Dyspnea Index focal score less than/equal to 6)
* Clinically stable as defined by no changes in medication dosage or frequency of administration with no exacerbations or hospital admissions in the preceding four weeks
* Males or females greater than 40 years of age;
* A cigarette smoking history of at least 20 pack-years
* Able to perform all study procedures and sign informed consent

Exclusion Criteria:

* History of asthma, atopy or nasal polyps
* Recent history of cardiovascular disease (< 1 year) or other significant disease that could contribute to dyspnea or exercise limitation
* Oxygen saturation less than 80% during exercise on room air

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2005-09; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
endurance time | 60 minutes post-inhalation
dyspnea | 60-minutes post-inhalation

CONTACTS AND LOCATIONS:
Overall Officials: Denis E O'Donnell, MD, Principal Investigator — Queen's University-Respiratory Investigation Unit
Locations (1):
- Respiratory Investigation Unit, Kingston, Ontario, Canada